CLINICAL TRIAL: NCT06120686
Title: Effect of Biofeedback Training on Cognitive and Motor Functions in Children With Intellectual Disabilities
Brief Title: Biofeedback Training's Impact on Cognitive and Motor Skills in Kids With Intellectual Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aleksandra Kiper (Other)
Responsible Party: Sponsor-Investigator, Aleksandra Kiper, Master of Physiotherapy, University of Rzeszow
Organization: University of Rzeszow (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023/07/48
Record Dates: First submitted 2023-10-14; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Intellectual Disability, Mild
Keywords: intellectual disability; cognitive function; motor function; training; rehabilitation; biofeedback
MeSH Terms: conditions — Intellectual Disability; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: random selection to two groups (study group and control group)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biofeedback-based therapy (BBT) (Experimental): study group - implementing the conventional therapy program supplemented additionally by training with visual and auditory biofeedback on a dynamic balance platform
  Interventions: Other: Biofeedback method; Other: Conventional therapy program
- conventional therapy program (CT) (Other): control group - implementing only the conventional therapy program
  Interventions: Other: Conventional therapy program

INTERVENTIONS:
Other: Biofeedback method — Study group - implementing a conventional therapy program supplemented additionally with visual and auditory biofeedback training on a dynamic balance platform
  Other Names: Conventional therapy program
  Arms: biofeedback-based therapy (BBT)
Other: Conventional therapy program — Control group - rehabilitation management aimed at improving cognitive and motor functions in children with mild intellectual disabilities.

SUMMARY:
The expected outcome of the study is to confirm or reject the hypothesis that traditional rehabilitation in combined with biofeedback training produces better results in improving motor and cognitive functions, relative to conventional rehabilitation.

In addition, the result of the study will be a protocol for dealing with school-aged children school-age children with impaired motor functions associated with impaired cognitive functions.

The developed material, will be a practical addition to therapeutic programs, Particularly useful in the work of psychological and pedagogical clinics, in offices of rehabilitation and sensory integration offices, or centers implementing early childhood development supporting child development.

DETAILED DESCRIPTION:
In accordance with the study design, children with intellectual disabilities who will participate in a 3-week rehabilitation program will be eligible for the study.

The research will be a single-center study. The research will be conducted at the St. Hedwig the Queen Regional Hospital No. 2, Lwowska 60, 35-301 Rzeszów - Department of Child Neurology and Pediatrics.

Number of subjects included in the study: The planned group size is 60 people (30 people - study group, 30 people - control group). The given population was calculated on the basis of the sampling calculator " PLUS module " Statistica 13.3 software, taking into account the following parameters: fraction size, confidence level, maximum error.

For the study of the effect of biofeedback training on cognitive and motor function in children with intellectual disabilities, there is no need to recruit healthy participants to the control group.

Prior to the actual study, a pilot study will be conducted on a smaller group of test subjects. After taking into account the eligibility criteria, the subjects will be assigned, on the basis of random selection random assignment, to two groups: the study group - implementing the conventional therapy program supplemented additionally with visual and auditory biofeedback training on a dynamic balance platform, the control - implementing only the conventional therapy program.

Respondents from both groups will participate in a 3-week therapy program, under the same conditions using the same measuring instruments. All participants will be informed about the purpose and conduct of the study and, after consenting to the study, will be qualified for the study proper. The participation of the child called "Minor" in this study depends solely on the parent or legal guardian's expression of consent by signing the Informed Consent Form after reading the information presented information about the study being conducted.

The examination will be performed twice, the initial one before the start of therapy, and the control one after the 3-week rehabilitation program has been completed. The following tools will be used to evaluate the effects of rehabilitation: AMTI dynamography platform, Romberg Test, Up and Go Test - assessment of static and dynanmic balance, ZEBRIS computer system - assessment of posture, HEG Biofeedback (hemoencephalography) - assessment of concentration and attention, AVLT (AuditoryVerbal Lerning Test), Bourdon-Wiersma Test - assessment of cognitive functions, Southern California Sensory Integration Test - assessment of sensory function, Box and Block Test, dynamometer - assessment of hand function, Eurofit Special Test - assessment of physical fitness, PedsQLTM Pediatric Quality of Life Questionnaire - assessment of quality of life, Barthel Scale - assessment of functional ability.

The examination time for one participant will be 1.5 hours. A period of 12 months is planned for recruitment and examination of participants.

The planned study does not involve any risks and possible health hazards for the participants examination. The conducted examination will be completely painless and non-invasive with dignity and principles of intimacy for each patient. The examination will be conducted using measuring devices certified and approved for use within the framework of scientific research in the field of rehabilitation.

The expected outcome of the study is to confirm or reject the hypothesis that traditional rehabilitation combined with biofeedback training produces better results in improving motor and cognitive functions, compared to conventional rehabilitation.

Description of benefits to study participants:

Improved motor and cognitive functions of children with intellectual disabilities, protocol rehabilitation management for children with intellectual disabilities.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed mild intellectual disability,
* age 7-12 years,
* current health status allowing the child to participate in the study and participate in the rehabilitation program,
* informed voluntary consent of parents and/or legal guardians to participate in the study.

Exclusion Criteria:

* diagnosed intellectual disability of severe and profound degree,
* cognitive deficits impairing the ability to understand and follow instructions,
* age below 7 or above 12 years,
* coexistence of autism, Down syndrome, cerebral palsy, muscular dystrophy and neurological disorders, such as epilepsy or brain damage,
* the presence of comorbidities such as rheumatic, orthopedic, oncological or cardiac diseases that may affect the subject's motor impairment.
* the lack of informed voluntary consent from parents and/or legal guardians to participate in the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of static and dynamic balance using the AMTI platform | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program.
  AMTI platform use is to assess balance ability.
Posture assessment using the computer-based ZEBRIS system | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program.
  Zebris device allows non-invasive assessment of the shape of the curvature of the spine and parameters that determine postural disorders. The ZEBRIS system consists of a measuring unit, a system of micro-sensors and an ultrasonic pointer, with which topographic points are scanned from the skeleton and then processed in a computer program in the form of a report containing numerical data specifying lengths, angles and degrees for each parameter, as well as graphs and figures of the spinal line.
Assessment of concentration and attention with HEG Biofeedback (hemoencephalography) | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program.
  Hemoencephalography (HEG) is a method of monitoring changes in frontal cerebral blood circulation and oxygenation. HEG biofeedback is a method based on the use of near-infrared technology to measure cerebral hemodynamics.
  A sensor armband is placed on the head in the area where reduced blood oxygenation is noted, and then emits into the brain, two beams of light at different frequencies. This allows us to check the oxygen saturation in a particular area of the brain in real time. The signal is returned to the computer screen, and the trainer tries to increase it. HEG biofeedback training involves stimulating neurons in the frontal lobes of the brain.

SECONDARY OUTCOMES:
Assessment of functional by Barthel Scale | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program.
  Based on the scores assigned the patient's condition is described in the following way: I. 86-100 points - "slight" dependency; II. 21- 85 points - "moderately severe" dependency; III. 0 - 20 points - "severe" dependency.
  ability
Quality of life assessment using the PedsQLTM Pediatric Quality of Life Questionnaire | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program
  The PedsQL is based on a modular approach to measuring health-related quality of life and consists of a 15-item core measure of global health-related quality of life .
Assessment of cognitive function using the AVLT test | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program
  Involves five sequential presentations of a 15-word list.
Assessment of cognitive function using the Bourdon-Wiersma test | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program
  The Bourdon test is an approach to measuring focus and attention that requires the test taker to detect and cross out specific characters in a set of letters.
Manual skills, assessed with Box and Blocks test | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program
  The test uses a wooden box, divided into two equal parts by a partition, as well as 150 blocks. The subject moves as many blocks as possible from one part of the box to the other during 60 seconds.
Romberg test | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program
  The Romberg test is used to assess static balance. The test involves standing with your feet together and your arms at your side or crossed in front of you. Part of the test is with your eyes open, and the second part is with your eyes closed.
TUG test | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program
  In the TUG test subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again.
Southern California Sensory Integration Test - Bilateral Motor Coordination | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program
  This test gives information about the motor activity of both sides of the body, sense of rhythm and sequence.
Southern California Sensory Integration Test - Crossing the Body's Midline | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program
  This test gives information about the rate and quality of cooperation between the brain hemispheres.
Southern California Sensory Integration Test - Graphesthesia | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program
  This test gives information about the ability to visualize tactile stimuli from the top of the hand area and visuomotor coordination.
Southern California Sensory Integration Test - Differentiating Right from Left | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program
  This test gives information about distinguishing the sides of the body.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rzeszów, Rzeszów, Poland